CLINICAL TRIAL: NCT00278096
Title: Randomised Controlled Trial of Unsolicited Occupational Therapy in Community-Dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUMC P 92/99; NWO014-91-006
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2006-01-18 (Estimated); Status verified 2006-01

CONDITIONS: Disability; Occupational Therapy
Keywords: disability; occupational therapy
MeSH Terms: interventions — Occupational Therapy

INTERVENTIONS:
Behavioral: occupational therapy

SUMMARY:
In this study we aim to assess whether unsolicited occupational therapy compared to no therapy can decelerate the increase in disability in high-risk elderly.

DETAILED DESCRIPTION:
Community-dwelling elderly, and particularly the oldest old, are generally viewed as highly susceptible to the 'inverse care law'. That is, those in greatest need for preventive assessment and surveillance have the highest potential benefit but are most likely to be missed. Hence, active case-finding and close follow-up might be an important strategy for maintaining the health, independence, and well-being of very elderly people who are at a particularly high risk.

In this study we aim to assess whether unsolicited occupational therapy compared to no therapy can decelerate the increase in disability in high-risk elderly. Subjects in the intervention group will be visited by an occupational therapist who provides training and education about assistive devices that are already present and will give recommendations and information about procedures, possibilities, and costs of assistive devices and community-based services. Control subjects will not be visited by an occupational therapist.

The primary outcome measure of the trial will be the score on the Groningen Activity Restriction Scale (GARS). Secondary outcome measures will be well-being and feelings of loneliness.

ELIGIBILITY:
Inclusion Criteria:

* age 85 years
* living independently
* MMSE score > 18 points

Exclusion Criteria:

* none

Ages: 85 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400
Dates: Start 2000-03; Study Completion 2004-05

PRIMARY OUTCOMES:
Score on the Groningen Activity Restriction Scale (GARS)

SECONDARY OUTCOMES:
Well-being and feelings of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Anton JM de Craen, PhD, Principal Investigator — Leiden University Medical Center